CLINICAL TRIAL: NCT03868462
Title: Optos P200TE Agreement and Precision Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Optos, PLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPT1029
Record Dates: First submitted 2019-03-02; First posted 2019-03-11 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Retinal Disease; Glaucoma
MeSH Terms: conditions — Retinal Diseases; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Optical Coherence Tomography (OCT) (Other)
  Interventions: Device: Optos P200TE; Device: Predicate Device

INTERVENTIONS:
Device: Optos P200TE — The P200TE Ophthalmoscope provides widefield Scanning Laser Ophthalmoscope (SLO) fundus imaging and Optical Coherence Tomography (OCT) imaging in one device.
Device: Predicate Device — The predicate device is an optical coherence tomography system intended for in vivo imaging, axial cross-sectional, three-dimensional imaging and measurement of anterior and posterior ocular structures.

SUMMARY:
This study is a prospective comparative, randomized, single center study to assess agreement and precision of the Optos P200TE in comparison to the predicate device in normal subjects, subjects with glaucoma, and subjects with retinal disease.

ELIGIBILITY:
Inclusion Criteria for Normal Group

1. Subjects 22 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects with normal eye examinations in both eyes on the date of the study visit as observed with a 90 diopter lens
4. BCVA 20/40 or better (each eye) on the date of the study visit

   Exclusion Criteria for Normal Group
5. Subjects unable to tolerate ophthalmic imaging
6. Subjects with ocular media not sufficiently clear to obtain acceptable OCT images in either eye
7. Presence of any ocular pathology except for cataract in either eye
8. History of leukemia, dementia or multiple sclerosis

   Inclusion Criteria for Glaucoma Group
9. Subjects 22 years of age or older on the date of informed consent
10. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
11. BCVA 20/40 or better in the study eye
12. History of Visual field defects within the previous six (6) months from the study visit or measured the day of the study visit consistent with glaucomatous optic nerve damage with at least one of the following two findings:

    1. On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level;
    2. Glaucoma hemi-field test "outside normal limits."
13. Glaucomatous optic nerve damage as evidenced by any of the following optic disc or retinal nerve fiber layer structural abnormalities:

    1. Diffuse thinning, focal narrowing, or notching of the neuroretinal rim, especially at the inferior or superior poles with or without disc hemorrhage;
    2. Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue

    Exclusion Criteria for Glaucoma Group
14. Subjects unable to tolerate ophthalmic imaging
15. Subjects with ocular media not sufficiently clear to obtain acceptable OCT images in the study eye
16. No reliable Humphrey Field Analyzer (HFA) visual field (24-2 Sita Standard, white on white) result within 6 months of the study visit, defined as fixation losses > 33% or false positives > 33%, or false negatives > 33% in the study eye
17. Presence of any ocular pathology except glaucoma in the study eye
18. History of leukemia, dementia or multiple sclerosis

    Inclusion Criteria for Retina Disease Group
19. Subjects 22 years of age or older on the date of informed consent
20. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
21. Subjects presenting at the site with retinal disease
22. BCVA 20/400 or better in the study eye
23. Diagnosis of some type of retinal pathology by investigator, may include, but not limited to: Macular Degeneration (including patients with drusen and geographic atropy and choroidal neovascularization), Diabetic Macular Edema, Diabetic Retinopathy, Macular Hole, Epiretinal Membrane, Central Serous Retinopathy and others

    Exclusion Criteria for Retinal Disease Group
24. Subjects unable to tolerate ophthalmic imaging
25. Subject with ocular media not sufficiently clear to obtain acceptable OCT images in the study eye
26. Presence of glaucoma or any ocular pathology other than a retinal pathology (e.g., cornea pathology) in the study eye as determined by self-report and/or investigator assessment at the study visit;
27. History of leukemia, dementia or multiple sclerosis

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Limit of Agreement (LOA) between the Optos P200TE and predicate device measurements of full retinal thickness (μm). | At the end of Visit 1 or optional Visit 2 (each visit is 1 day)
Limit of Agreement (LOA) between the Optos P200TE and predicate device measurements of retinal nerve fiber layer thickness (μm). | At the end of Visit 1 or optional Visit 2 (each visit is 1 day)
Limit of Agreement (LOA) between the Optos P200TE and predicate device measurements of ganglion cell complex thickness (μm). | At the end of Visit 1 or optional Visit 2 (each visit is 1 day)
Limit of Agreement (LOA) between the Optos P200TE and predicate device measurements of optic disc (area, volume, cup-to-disc ratio). | At the end of Visit 1 or optional Visit 2 (each visit is 1 day)
Precision between the Optos P200TE and predicate device measurements of full retinal thickness. | At the end of Visit 1 or optional Visit 2 (each visit is 1 day)
Precision between the Optos P200TE and predicate device measurements of retinal nerve fiber layer thickness. | At the end of Visit 1 or optional Visit 2 (each visit is 1 day)
Precision between the Optos P200TE and predicate device measurements of ganglion cell complex thickness. | At the end of Visit 1 or optional Visit 2 (each visit is 1 day)
Precision between the Optos P200TE and predicate device measurements of optic disc (area, volume, cup-to-disc ratio). | At the end of Visit 1 or optional Visit 2 (each visit is 1 day)
Precision of the P200TE for the super pixel grid measurements of the full retinal thickness. | At the end of Visit 1 or optional Visit 2 (each visit is 1 day)
Precision of the P200TE for the super pixel grid measurements of the RNFL thickness. | At the end of Visit 1 or optional Visit 2 (each visit is 1 day)
Precision of the P200TE for the super pixel grid measurements of GCC thickness. | At the end of Visit 1 or optional Visit 2 (each visit is 1 day)

CONTACTS AND LOCATIONS:
Locations (1):
- New England Retina Consultants, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No